CLINICAL TRIAL: NCT06781658
Title: Rehab in Mild DCM: Study Protocol for a Feasibility Randomised Controlled Trial to Compare the Effectiveness of a Structured Rehabilitation Intervention to Clinical Surveillance in People With Mild Stable Degenerative Cervical Myelopathy.
Brief Title: Rehab in Mild Stable DCM: Feasibility RCT Comparing Structured Rehabilitation to Clinical Surveillance
Acronym: RehabmildDCM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-172
Record Dates: First submitted 2025-01-06; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Degenerative Cervical Myelopathy
Keywords: Degenerative cervical myelopathy; Mild DCM; Rehabilitation; clinical Surveillance; Feasibility RCT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Every participant will have a unique identifier. The outcome assessors will be blinded to group allocation. Clinicians delivering the interventions and trial participants will not be blinded to group allocations due to the nature of the intervention (56). Participants will be asked in advance of attending for their 12 week follow up not to disclose their group allocation with the outcome assessor. Data analysts will be blinded to group allocation. Unblinding will only occur in exceptional circumstances when knowledge of the group allocation is essential for further management of the participant (57).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured rehabilitation intervention (Experimental): The SRI will include education, a physical activity behavioural change intervention, cervical range of motion exercises, neck, upper limb and scapular strengthening exercises and task specific hand function training.
  Interventions: Other: Structured rehabilitation intervention
- Clinical surveillance (Active Comparator): Participants assigned to the clinical surveillance control group will be invited to attend a single, one to one education session which will be supplemented with a written patient information booklet after which they will be scheduled for a 12 week follow up.
  Interventions: Other: Clinical Surveillance

INTERVENTIONS:
Other: Structured rehabilitation intervention — Participants will be prescribed a multi-component SRI which will include education, cervical range of motion exercises, progressive neck strengthening exercises, individualised scapular and upper limb strengthening, task specific hand function training and a physical activity behavioural change intervention. The TIDieR checklist has been used to provide a comprehensive description of this complex intervention. (17).
  Arms: Structured rehabilitation intervention
Other: Clinical Surveillance — Participants assigned to the clinical surveillance control group will be invited to attend a single, one to one education session which will be supplemented with a written patient information booklet after which they will be scheduled for a 12 week follow up.
  Arms: Clinical surveillance

SUMMARY:
The goal of this feasibility RCT is to establish the feasibility of undertaking a RCT investigating the effectiveness of a multi component structured rehabilitation intervention aiming at reducing physical disability in people with mild stable Degenerative Cervical Myelopathy. The main question it will answer are what is the incidence of mild stable DCM in the neurosurgical OPD clinics, what is the eligibility rate and participate rate of those eligible. It will also investigate the acceptability of the intervention to both participants and clinicians and participant retention.

Researchers will compare a structured rehabilitation intervention to clinical surveillance. The structured rehabilitation intervention will include education, a physical activity behavioural change intervention, cervical range of motion exercises, neck, upper limb and scapular strengthening exercises and task specific hand function training.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of DCM (Clinical symptom of DCM +/- Upper motor neuron sign + imaging evidence of cervical cord compression). Diagnosis will be confirmed by a consultant neurosurgeon (19).

  * Modified Japanese Orthopaedic assessment (mJOA) score of 15-17, indicating mild DCM. The mJOA is a clinician administered validated measure of DCM severity (20)
  * Adequate comprehension of English to understand the purpose of the study and give written informed consent

Exclusion Criteria:

* Patient or surgeon preference for urgent surgical decompression for progressive DCM, motor radiculopathy or severe unrelenting radicular arm pain or significant risk factors for progression including co-existing cervical radiculopathy and circumferential cord compression.

  * Diagnosis of other neurological condition that could confound assessment.
  * Involvement in another clinical study or trial
  * Pregnancy
  * If the participant is unable to commit to a 12-week programme of up to 10 sessions of supervised rehabilitation and participating in a regular home exercise programme for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-13 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of mild stable DCM | Baseline
  Number of people with mild stable DCM during the study period/ number of NP seen.
Number of people with mild stable DCM who are willing to participate but do not reach the eligibility criteria | Baseline
  The number of people with mild stable DCM over the study period- the number of people with mild stable DCM who are eligible to participate in the study.
Participant recruitment rate | Baseline
  The number of participants recruited per month
Participant adherence to the intervention | 12 weeks
  The number of scheduled sessions attended by the participants.
Clinician adherence to the intervention | 12 weeks
  The number of core intervention components included in each treatment session
Acceptability of the intervention to the participants and clinicians | 12 weeks
  Semi-structured interviews
Burden of measurement tool completion | 12 weeks
  Semi structured interview
Participant retention rate | 12 weeks
  Loss to follow up rate and reasons for loss to follow up

SECONDARY OUTCOMES:
Physical component score of the short form (SF) 36 | Baseline and 12 weeks
  Physical functioning
Modified Japanese Orthopaedic association index (mJOA) | Baseline and 12 weeks
  Myelopathy severity scale
Neck disability index | Baseline and 12 weeks
  Neck pain related disability
Spinal adverse events severity scale | 12 weeks
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ciaran Bolger, MD PhD, Principal Investigator — Royal College of Surgeons
Locations (1):
- Beaumont Hospital, Dublin, Ireland